CLINICAL TRIAL: NCT05802381
Title: the Safety and Effectiveness of Protein Supplements on Cancer Patients With Nutritional Risk and Malnutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: protein-malnutrition-cancer
Record Dates: First submitted 2023-03-27; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Malnutrition
Keywords: protein; malnutrition; nutritional risk; cancer
MeSH Terms: conditions — Neoplasms; Malnutrition | interventions — Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- protein supplements (Experimental): This group will receive dietary guidance and protein supplements for 3 months
  Interventions: Dietary Supplement: protein supplement; Behavioral: nutrition counseling
- dietary guidance (Other): this group will receive dietary guidance for 3 months
  Interventions: Behavioral: nutrition counseling

INTERVENTIONS:
Dietary Supplement: protein supplement — 20 gram protein supplement per day
  Other Names: protein
  Arms: protein supplements
Behavioral: nutrition counseling — nutrition counseling for guidance of food intake

SUMMARY:
Nutritional risk and malnutrition is common in cancer patients, which is one of the significant factors affecting the overall survival, toxicity during anticancer treatment, and quality of life among patients with cancer. Previous studies have shown that the increased protein intake can stimulate muscle synthesis, and improve muscle mass, strength, function, overall survival, and quality of life. The current study is going to investigate the effectiveness and safety of protein supplements on patients with cancer, in order to provide a reference for further nutrition treatment.

DETAILED DESCRIPTION:
An anticipated total of 100 participants will randomly assigned to receive either a 20-gram protein supplement per day or nutrition counseling to increase the protein intake. there will be a total of 3 study visits, and dietary assessment and blood sample collection will occur at every study visit. Intention-to-treat analysis (ITT) and per-protocol analysis (PP) will be used in statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Age>=18years old;

  * Initial treatment patients with lung/gastrointestinal/esophageal cancer
  * Patients with nutritional risk (NRS-2002≥3) ;
  * Patients are able to provide written informed consent.

Exclusion Criteria:

* • People who are allergic to whey protein.

  * Participants received any drugs or supplements known to influence the outcomes, such as protein powder, anabolic steroids, or glucocorticoids before the 3 months preceding the study.
  * Participants with gastrointestinal bleeding or intestinal obstruction, or any contraindication for oral intake
  * Concurrent severe cardiac disease, liver and renal failure, which may significantly interfere with study compliance.
  * Participants with electronic or mental device.
  * Women in pregnancy or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
blood toxicity | 6 month
  blood toxicity based on Common Terminology Criteria for Adverse Events (CTCAE)
nutritional risk | 6 months
  nutritional risk based on nutrition risk screening-2002 (NRS-2002)
malnutrition | 6 months
  malnutrition assessment based on Global Leadership Initiative on Malnutrition (GLIM)

SECONDARY OUTCOMES:
phase angle (PA) | 6 month
  phase angle (PA) assessed by multi-Bioelectric Impedance Analysis (m-BIA)
weight | 6 month
  weight change during the study
dose limitation | 6 months
  dose limitation

CONTACTS AND LOCATIONS:
Overall Officials: Kang Yu, MD, Study Director — Peking Union Medical College Hospital; Fang Wang, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No